CLINICAL TRIAL: NCT03271931
Title: Using Active Choice in the EHR to Promote Cardiologists to Prescribe Evidence-Based Statin Therapy
Brief Title: Active Choice in the EHR to Promote Statin Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 827983
Record Dates: First submitted 2017-09-01; First posted 2017-09-05 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual care (No Intervention): Cardiologists in this arm will receive no interventions and will act as usual care
- Active choice (Experimental): Cardiologists in this arm will be exposed to an active choice intervention through the electronic health record (EHR) using an alert to prompt recommendations for statin therapy for patients not on guideline-based therapy. Cardiologists will be have to make an active choice to prescribe a statin at the recommended dose or not.
  Interventions: Behavioral: Active choice
- Passive choice (Experimental): Cardiologists in this arm will be exposed to a passive choice alert within the EHR, using the same evidence-based guidelines as in the active choice arm. The passive alert will not block clinician workflow and instead will be available in the background for the cardiologist to open and then use to make a prescribing decision.
  Interventions: Behavioral: Passive choice

INTERVENTIONS:
Behavioral: Active choice — EHR alert prompting cardiologists to make an active choice to prescribe a statin or not.
  Arms: Active choice
Behavioral: Passive choice — EHR passive alert to cardiologists about prescribing a statin
  Arms: Passive choice

SUMMARY:
Cardiovascular (CV) events are the leading cause of mortality in the United States. Statins have been demonstrated to be an effective tool for reducing CV events and mortality, but statins are often either not prescribed or under-prescribed for patients that meet evidence-based guidelines. In this study, we will evaluate a health system initiative using active and passive choice prompts in the electronic health record to prompt cardiologists to prescribe evidence-based statin therapy. In partnership with the health system, this will be conducted as a randomized, controlled trial to evaluate its effect.

DETAILED DESCRIPTION:
This study will use a randomized, controlled trial to evaluate a health system initiative. Cardiologists randomly assigned to the control arm will receive no interventions. For cardiologists randomly assigned to the active choice intervention, the electronic health record will be used to prompt cardiologists to initiate or change statin therapy for patients not on evidenced-based guidelines based on the 2013 American College of Cardiology / American Heart Association (ACC/AHA) and the National Lipid Association (NLA) through a "best practice alert" in Epic which appears on the screen and forces a decision before the clinician can move on. For cardiologists randomly assigned to the passive choice intervention, the electronic health record will be used to create a passive alert using the same evidence-based guidelines. The passive alert will not block clinician workflow and instead will be available in the background for the cardiologist to open and then use to make a prescribing decision. The intervention period will be 6 months in duration.

ELIGIBILITY:
Inclusion Criteria:

* Have a cardiologist at the University of Pennsylvania Health System
* Meets 2013 ACC/AHA or NLA guidelines for statin prescription

Exclusion Criteria:

* Allergy to statins
* Severe renal insufficiency defined as glomerular filtration rate (GFR) less than 30 mL/min or on dialysis
* Adverse reaction to statins including a) myopathy, b)rhabdomyolysis, c)hepatitis
* Pregnant
* On a PCSK9 Inhibitor medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23066 (Actual)
Dates: Start 2018-09-24 (Actual); Primary Completion 2019-06-05 (Actual); Study Completion 2019-06-05 (Actual)

PRIMARY OUTCOMES:
Change in the percent of eligible patients prescribed statin therapy at a dose that meets evidence-based guidelines | 6 Months
  Among patients not on guideline-based statin dosages, the percent that are prescribed guideline-based therapy at appropriate dose.

SECONDARY OUTCOMES:
Change in percentage of eligible patients prescribed a statin, at any dose. | 6 Months
  Among patients not on a statin, the percent that are prescribed guideline-based therapy, at any dose.

CONTACTS AND LOCATIONS:
Overall Officials: Mitesh Patel, MD, MBA, MS, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Adusumalli S, Westover JE, Jacoby DS, Small DS, VanZandbergen C, Chen J, Cavella AM, Pepe R, Rareshide CAL, Snider CK, Volpp KG, Asch DA, Patel MS. Effect of Passive Choice and Active Choice Interventions in the Electronic Health Record to Cardiologists on Statin Prescribing: A Cluster Randomized Clinical Trial. JAMA Cardiol. 2021 Jan 1;6(1):40-48. doi: 10.1001/jamacardio.2020.4730. PMID 33031534